CLINICAL TRIAL: NCT01078623
Title: Efficacy, Safety and Tolerability of Two Fixed-Dose Combinations of Aclidinium Bromide With Two Doses of Formoterol Fumarate Compared With Aclidinium Bromide, Formoterol Fumarate and Placebo All Administered Twice Daily in Stable, Moderate to Severe Chronic Obstructive Pulmonary Disease Patients.
Brief Title: Efficacy and Safety of Two Fixed Dose Combinations of Aclidinium Bromide With Formoterol Fumarate
Acronym: ALIGHT-COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/40464/26
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Bronchitis; Chronic; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Bronchiolitis Obliterans Syndrome; Emphysema | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Formoterol 12 μg (Active Comparator): Formoterol fumarate 12 μg twice daily
  Interventions: Drug: Formoterol 12 μg
- Placebo (Placebo Comparator): Placebo twice daily
  Interventions: Drug: Placebo
- Aclidinium 200 μg / formoterol 12 μg (Experimental): Aclidinium bromide 200 μg + formoterol fumarate 12 μg fixed dose combination (FDC) twice daily
  Interventions: Drug: Aclidinium 200 μg / formoterol 12 μg
- Aclidinium 200 μg / formoterol 6 μg (Experimental): Aclidinium bromide 200 μg + formoterol fumarate 6 μg fixed dose combination (FDC) twice daily
  Interventions: Drug: Aclidinium 200 μg / Formoterol 6 μg
- Aclidinium 200 μg (Experimental): Aclidinium bromide 200 μg twice daily
  Interventions: Drug: Aclidinium 200 μg

INTERVENTIONS:
Drug: Aclidinium 200 μg / formoterol 12 μg — Aclidinium bromide 200 μg + formoterol fumarate 12 μg fixed dose combination (FDC) twice daily
  Arms: Aclidinium 200 μg / formoterol 12 μg
Drug: Placebo — Placebo control twice daily
  Arms: Placebo
Drug: Formoterol 12 μg — Formoterol fumarate 12 μg twice daily
  Arms: Formoterol 12 μg
Drug: Aclidinium 200 μg — Aclidinium bromide 200 μg twice daily
  Arms: Aclidinium 200 μg
Drug: Aclidinium 200 μg / Formoterol 6 μg — Aclidinium bromide 200 μg + formoterol fumarate 6 μg fixed dose combination (FDC) twice daily
  Arms: Aclidinium 200 μg / formoterol 6 μg

SUMMARY:
The purpose of this multicenter, dose-ranging study is to compare two Fixed-Dose Combinations of aclidinium bromide and formoterol fumarate with placebo, aclidinium bromide and formoterol fumarate, all administered BID in patients with stable, moderate to severe COPD.

Every treatment period is 14-days long and there is a 7-days wash-out period in between them. The trial starts with a run in phase of 10 to 17-days duration and it ends up with a follow up contact 14-days after last treatment dose.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or non-pregnant, non-lactating female aged between 40 and 80 years old, both inclusive.
2. Patient with a clinical diagnosis of stable moderate to severe COPD according to the GOLD classification
3. Current, or ex-cigarette smoker with a smoking history of at least 10 pack-years.
4. Patient whose FEV1 at the Screening Visit measured between 10-15 minutes post inhalation of 400 mcg of salbutamol is 30% FEV1 <80% of the predicted normal value (i.e., 100 x Post-salbutamol < FEV1/ Predicted FEV1 must be < 80% and ≥ 30%).
5. Patient whose FEV1/FVC at the Screening Visit measured between 10-15 minutes post inhalation of 400 mcg of salbutamol is < 70% (i.e., 100 x Post-salbutamol FEV1 /FVC < 70%).
6. Patient who is eligible and able to participate in the trial and who consent to do so in writing after the purpose and nature of the investigation have been explained.
7. Patient whose COPD symptoms and FEV1 values at the time of randomisation are stable compared to the Screening Visit, according to the investigator's medical judgment

Exclusion Criteria:

1. History or current diagnosis of asthma or exercise-induced bronchospasm.
2. Clinically significant respiratory conditions at the time of Inform Consent signature
3. Hospitalisation due to COPD exacerbation within the previous 3 months.
4. Signs of a COPD exacerbation or respiratory infection (including the upper respiratory tract) within the previous 6 weeks.
5. Patient who has a resting systolic blood pressure ≥ 200 mmHg, a resting diastolic blood pressure ≥ 120 mmHg or a resting heart rate ≥ 105 bpm at screening visit.
6. Clinically significant cardiovascular conditions
7. Presence of symptomatic prostatic hypertrophy and/or bladder neck obstruction.
8. Presence of narrow-angle glaucoma.
9. QTc [calculated according to Bazett's formulae (QTc=QT/RR1/2) above 470 milliseconds in the ECG performed at Screening Visit,
10. Patient who does not maintain regular day/night, waking/sleeping cycles

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (10):
- Czechia (4):
  - Research Site, Bucuresti
  - Research Site, Constanta
  - Research Site, Iasi
  - Research Site, Tg Mures
- Romania (6):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Timișoara

REFERENCES:
- See also: Almirall Corporate Website — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3971&filename=Synopsis%20m-40464-26-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a total of 28 sites (4 sites in Czech Republic, 5 sites in Germany, 3 sites in Hungary, 4 sites in Poland and 12 sites in Romania)
  The first patient was screened in February 2010 and the last patient visit was in September 2010
Pre-assignment Details: A total of 176 patients were screened of whom 135 were assessed as eligible and were randomized into the study
  There were 41 screen failures, the main reason being non-fulfilment of inclusion/exclusion criteria
Groups:
- Sequence 1: FDC 200/6 μg - FDC 200/12 μg - Aclidinium 200 μg - Formoterol 12 μg
- Sequence 2: FDC 200/12 - Aclidinium 200 - Formoterol 12 - Placebo
- Sequence 3: Aclidinium 200 - Formoterol 12 - Placebo - FDC 200/6
- Sequence 4: Formoterol 12 - Placebo - FDC 200/6 - FDC 200/12
- Sequence 5: Placebo - FDC 200/6 - FDC 200/12 - Aclidinium 200
- Sequence 6: FDC 200/6 - Aclidinium 200 - Placebo - FDC 200/12
- Sequence 7: FDC 200/12 - Formoterol 12 - FDC 200/6 - Aclidinium 200
- Sequence 8: Aclidinium 200 - Placebo - FDC 200/12 - Formoterol 12
- Sequence 9: Formoterol 12 - FDC 200/6 - Aclidinium 200 - Placebo
- Sequence 10: Placebo - FDC 200/12 - Formoterol 12 - FDC 200/6
- Sequence 11: FDC 200/6 - Formoterol 12 - FDC 200/12 - Placebo
- Sequence 12: FDC 200/12 - Placebo - Aclidinium 200 - FDC 200/6
- Sequence 13: Aclidinium 200 - FDC 200/6 - Formoterol 12 - FDC 200/12
- Sequence 14: Formoterol 12 - FDC 200/12 - Placebo - Aclidinium 200
- Sequence 15: Placebo - Aclidinium 200 - FDC 200/6 - Formoterol 12
- Sequence 16: FDC 200/6 - Placebo - Formoterol 12 - Aclidinium 200
- Sequence 17: FDC 200/12 - FDC 200/6 - Placebo - Formoterol 12
- Sequence 18: Aclidinium 200 - FDC 200/12 - FDC 200/6 - Placebo
- Sequence 19: Formoterol 12 - Aclidinium 200 - FDC 200/12 - FDC 200/6
- Sequence 20: Placebo - Formoterol 12 - Aclidinium 200 - FDC 200/12
Period: Treatment Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 6 | 6 | 7 | 6 | 7 | 6 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7
Completed | 5 | 5 | 6 | 6 | 7 | 5 | 6 | 6 | 5 | 6 | 6 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 5 | 5 | 6 | 6 | 7 | 5 | 6 | 6 | 5 | 6 | 6 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 7
Completed | 5 | 5 | 6 | 6 | 7 | 4 | 5 | 6 | 5 | 6 | 6 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 5 | 5 | 6 | 6 | 7 | 4 | 5 | 6 | 5 | 6 | 6 | 7 | 7 | 7 | 7 | 7 | 7 | 7 | 6 | 7
Completed | 5 | 5 | 6 | 6 | 6 | 4 | 5 | 6 | 5 | 6 | 6 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10 | Sequence 11 | Sequence 12 | Sequence 13 | Sequence 14 | Sequence 15 | Sequence 16 | Sequence 17 | Sequence 18 | Sequence 19 | Sequence 20
Started | 5 | 5 | 6 | 6 | 6 | 4 | 5 | 6 | 5 | 6 | 6 | 7 | 7 | 6 | 7 | 7 | 7 | 7 | 6 | 7
Completed | 5 | 5 | 5 | 6 | 6 | 4 | 5 | 6 | 5 | 6 | 6 | 7 | 7 | 6 | 7 | 6 | 7 | 7 | 6 | 7
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All patients randomized into the study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (7.93)
Gender [Count of Participants; unit: Participants]
  Female | 40
  Male | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve Over 12 Hours (AUC0-12h) After Morning Study Drug Administration at Day 14
Description: FEV1 was measured via spirometry: 2 sets of tests prior to morning dose separated by 30 minutes, and then 1 set at 30 minutes, 1, 2, 3, 4, 6, 8, 10 and 12 hours post-morning dose
Time Frame: 0 and 30 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post-morning dose at Day 14
Population: Intent to treat (ITT) population: all randomized patients who took at least 1 dose of study drug and had at least 1 baseline and 1 post-baseline assessment of value of FEV1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Aclidinium 200 μg / Formoterol 12 μg: Aclidinium bromide 200 μg + formoterol fumurate 12 μg fixed dose combination (FDC) twice daily
- Aclidinium 200 μg / Formoterol 6 μg: Aclidinium bromide 200 μg + formoterol fumurate 6 μg fixed dose combination (FDC) twice daily
- Formoterol 12 μg: Formoterol fumurate 12 μg twice daily
Arm/Group | Placebo | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg | Formoterol 12 μg
Number analyzed (Participants) | 97 | 99 | 100 | 96 | 99
Liters | -0.041 (0.021) | 0.180 (0.021) | 0.193 (0.021) | 0.139 (0.021) | 0.100 (0.021)
Statistical Analysis 1: Comparison: Placebo vs Aclidinium 200 μg / Formoterol 12 μg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, subject as random effect, and baseline values at each period as a covariate; Least squares mean difference = 0.221, 95% CI 2-sided [0.174 to 0.268], Standard Error of Mean 0.024
Statistical Analysis 2: Comparison: Placebo vs Aclidinium 200 μg / Formoterol 6 μg; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, subject as random effect, and baseline values at each period as a covariate; Least squares mean difference = 0.234, 95% CI 2-sided [0.186 to 0.281], Standard Error of Mean 0.024

2. Secondary Outcome: Change From Baseline in Morning Pre-dose FEV1 at Day 14
Description: FEV1 was measured via spirometry: 2 sets of tests prior to morning dose separated by 30 minutes
Time Frame: Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg | Formoterol 12 μg
Number analyzed (Participants) | 100 | 99 | 100 | 96 | 99
Liters | -0.059 (0.020) | 0.042 (0.020) | 0.067 (0.020) | 0.072 (0.020) | 0.027 (0.020)

3. Secondary Outcome: Change From Baseline in Morning Peak FEV1 at Day 14
Description: as for outcome 1
Time Frame: 0 and 30 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post-morning dose at Day 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg | Formoterol 12 μg
Number analyzed (Participants) | 100 | 99 | 100 | 96 | 99
Liters | 0.052 (0.023) | 0.335 (0.023) | 0.347 (0.023) | 0.255 (0.023) | 0.255 (0.023)

ADVERSE EVENTS:
Time Frame: Up to 14 days following last dose of the investigational medicinal product (given over 14±2 days of treatment per period, with 4 treatment periods per patient)
Arm/Group | Placebo | Aclidinium 200 μg / Formoterol 12 μg | Aclidinium 200 μg / Formoterol 6 μg | Aclidinium 200 μg | Formoterol 12 μg
Serious Adverse Events (participants affected / at risk) | 0/101 | 2/101 | 0/102 | 0/100 | 1/101
Other Adverse Events (participants affected / at risk) | 0/101 | 0/101 | 0/102 | 0/100 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Aclidinium 200 μg / Formoterol 12 μg (N=101) | Aclidinium 200 μg / Formoterol 6 μg (N=102) | Aclidinium 200 μg (N=100) | Formoterol 12 μg (N=101)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and/or presentation whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and sponsor